CLINICAL TRIAL: NCT06102473
Title: Effect of a Digital Educational Intervention About the Front of Package Labeling of Industrialized Foods and Beverages on the Selection and Purchase of Products in Mexican Caregivers and Schoolchildren.
Brief Title: Effect of an Educational Intervention About Front of Package Labeling in Children and Caregivers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diana Avila Montiel (Other)
Responsible Party: Sponsor-Investigator, Diana Avila Montiel, Researcher in Medical Science, Hospital Infantil de Mexico Federico Gomez
Organization: Hospital Infantil de Mexico Federico Gomez (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIM/2022/054
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity; Malnutrition, Child
Keywords: front-of-package; warning labeling; food selection; children; caregivers; nutritional education
MeSH Terms: conditions — Overweight; Obesity; Child Nutrition Disorders; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The dyads (children and caregivers), will receive general nutritional education and also receive guidance on the use of front-of-package warning labels and awareness about the impact of the consumption of processed and ultra-processed foods on health.
  Interventions: Other: Nutritional education
- Control Group (No Intervention): The dyads (children and caregivers), will receive general nutritional education.

INTERVENTIONS:
Other: Nutritional education — With prior authorization from the principals of the elementary schools, meetings will be held with parents to invite them to participate, and the aim, activities, and duration of the intervention will be explained to them. They will be invited to sign a consent and informed assent, clarifying that their participation is voluntary and they may not continue at any time they wish without affecting their activities at school.
  Other Names: Educational
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of a digital educational intervention of front-of-package warning labeling on the selection and purchase of food in elementary school children and their caregivers.

The main question it aims to answer is:

* What is the effect of a digital educational intervention on front-of-package warning labeling on food selection in children from primary schools in Mexico City, compared to a control group? Participants will be randomized into two groups.
* The control group, the dyads (caregiver-schoolchildren), will receive general nutritional education.
* The intervention group, will also receive guidance on reading labels and raise awareness about the impact of consuming processed or ultra-processed foods on health.

The intervention will be carried out through a web page with audiovisual material and all participants also will be asked to complete:

* Multiple-choice evaluation (5 questions) to ensure theoretical understanding of the topics
* Lunch register
* 24-hour dietary recall
* Survey of food habits and consumption
* Validated food preference questionnaire
* Anthropometric measurements (Weight, height, waist circumference, body mass index)
* Socioeconomic survey
* Participate in a simulated online selection and shopping of food and beverages.

To see if the digital educational intervention in the front of package warning labeling in children and caregivers will improve the selection and purchase of foods.

DETAILED DESCRIPTION:
Third, fourth, and fifth-grade elementary school students and their caregivers from 4 primary schools, two public and two private, in Mexico City, will participate. The schools will be chosen by simple random sampling. Schools will be randomized into two groups: intervention and control.

After approval from the directors of the primary schools, meetings will be held with parents to invite them to participate, they will be explained the objectives, activities, and duration of the intervention. They will be invited to sign a consent and informed assent, clarifying that their participation is voluntary and they may not continue at any time they wish without affecting their activities at school.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Third, 4th, and 5th grade students, both sexes, enrolled in the selected primary schools.
* Children with normal weight, overweight, and obesity.
* Children who sign the written informed consent.

Caregivers:

* Primary caregivers of any sex for children in 3rd, 4th, and 5th grade
* Caregivers with normal weight, overweight and obesity
* Parents who sign the written informed consent

Exclusion Criteria:

Caregivers and children:

* No Internet Access
* No computer or mobile devices
* Who are participating in a weight reduction program, with or without pharmacological treatment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 404 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Food and drink selection | 1 week before starting the intervention, 3 months and 6 months
  Percentage of products purchased by each participant in the virtual store, whose content indicates "high in calories", sugar, fat, and sodium" and also average content of these nutrients in 100 g of the products.
Energy and macronutrient intake | 1 week before starting the intervention, 3 months and 6 months
  Amount of Kcal consumed, saturated fat, trans fat, sodium, added sugar

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Klünder-Klünder, PhD, Study Director — Hospital Infantil de Mexico Federico Gomez

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Neal B, Crino M, Dunford E, Gao A, Greenland R, Li N, Ngai J, Ni Mhurchu C, Pettigrew S, Sacks G, Webster J, Wu JH. Effects of Different Types of Front-of-Pack Labelling Information on the Healthiness of Food Purchases-A Randomised Controlled Trial. Nutrients. 2017 Nov 24;9(12):1284. doi: 10.3390/nu9121284. PMID 29186803
- [Background] Machin L, Arrua A, Gimenez A, Curutchet MR, Martinez J, Ares G. Can nutritional information modify purchase of ultra-processed products? Results from a simulated online shopping experiment. Public Health Nutr. 2018 Jan;21(1):49-57. doi: 10.1017/S1368980017001185. Epub 2017 Jul 18. PMID 28716163
- [Background] Vanderlee L, Franco-Arellano B, Ahmed M, Oh A, Lou W, L'Abbe MR. The efficacy of 'high in' warning labels, health star and traffic light front-of-package labelling: an online randomised control trial. Public Health Nutr. 2021 Jan;24(1):62-74. doi: 10.1017/S1368980020003213. Epub 2020 Oct 6. PMID 33019950
- [Background] Vilaro MJ, Barnett TE, Mathews A, Pomeranz J, Curbow B. Income differences in social control of eating behaviors and food choice priorities among southern rural women in the US: A qualitative study. Appetite. 2016 Dec 1;107:604-612. doi: 10.1016/j.appet.2016.09.003. Epub 2016 Sep 7. PMID 27612560
- [Background] Arrua A, Curutchet MR, Rey N, Barreto P, Golovchenko N, Sellanes A, Velazco G, Winokur M, Gimenez A, Ares G. Impact of front-of-pack nutrition information and label design on children's choice of two snack foods: Comparison of warnings and the traffic-light system. Appetite. 2017 Sep 1;116:139-146. doi: 10.1016/j.appet.2017.04.012. Epub 2017 Apr 18. PMID 28428151
- [Background] Tarabashkina L, Quester P, Crouch R. Exploring the moderating effect of children's nutritional knowledge on the relationship between product evaluations and food choice. Soc Sci Med. 2016 Jan;149:145-52. doi: 10.1016/j.socscimed.2015.11.046. Epub 2015 Dec 8. PMID 26717561
- [Background] Palfreyman Z, Haycraft E, Meyer C. Parental modelling of eating behaviours: observational validation of the Parental Modelling of Eating Behaviours scale (PARM). Appetite. 2015 Mar;86:31-7. doi: 10.1016/j.appet.2014.08.008. Epub 2014 Aug 8. PMID 25111293
- [Background] Vilchis-Gil J, Galvan-Portillo M, Klunder-Klunder M, Cruz M, Flores-Huerta S. Food habits, physical activities and sedentary lifestyles of eutrophic and obese school children: a case-control study. BMC Public Health. 2015 Feb 11;15:124. doi: 10.1186/s12889-015-1491-1. PMID 25885348
- [Background] Rodriguez-Ramirez S, Mundo-Rosas V, Garcia-Guerra A, Shamah-Levy T. Dietary patterns are associated with overweight and obesity in Mexican school-age children. Arch Latinoam Nutr. 2011 Sep;61(3):270-8. PMID 22696895
- [Background] Hawkes C, Smith TG, Jewell J, Wardle J, Hammond RA, Friel S, Thow AM, Kain J. Smart food policies for obesity prevention. Lancet. 2015 Jun 13;385(9985):2410-21. doi: 10.1016/S0140-6736(14)61745-1. Epub 2015 Feb 19. PMID 25703109
- [Background] Monasta L, Batty GD, Macaluso A, Ronfani L, Lutje V, Bavcar A, van Lenthe FJ, Brug J, Cattaneo A. Interventions for the prevention of overweight and obesity in preschool children: a systematic review of randomized controlled trials. Obes Rev. 2011 May;12(5):e107-18. doi: 10.1111/j.1467-789X.2010.00774.x. PMID 20576004
- [Background] Walley AJ, Asher JE, Froguel P. The genetic contribution to non-syndromic human obesity. Nat Rev Genet. 2009 Jul;10(7):431-42. doi: 10.1038/nrg2594. PMID 19506576
- [Derived] Avila-Montiel D, Vilchis-Gil J, Miranda-Lora AL, Velazquez-Lopez L, Klunder-Klunder M. The Effects of an Educational Intervention About Front-of-Package Labeling on Food and Beverage Selection Among Children and Their Caregivers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 1;13:e54783. doi: 10.2196/54783. PMID 38557591
- See also: National Health Survey — https://insp.mx/produccion-editorial/novedades-editoriales/ensanut-2018-nacionales
- See also: Front of package labeling of food and beverages — https://www.gob.mx/promosalud/acciones-y-programas/etiquetado-de-alimentos